CLINICAL TRIAL: NCT05250141
Title: Bioavailability of a Formulation of Oseltamivir Phosphate 75 mg Tablets With Regards to the Reference Product
Brief Title: Bioavailability of Levodopa 250 mg and Carbidopa 25 mg With Regards to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP8813-01
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Levodopa; Carbidopa; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levodopa and Carbidopa Test Product (Experimental): Participants will receive one tablet of the test formulation containing Levodopa and Carbidopa 250 mg/ 25 mg. The tablet will be taken with water and in a fasting condition.
  Interventions: Drug: Levodopa 250mg and Carbidopa 25mg Test Drug tablet
- Levodopa and Carbidopa Referent Product (Experimental): Participants will receive one tablet of the marketed reference containing Levodopa and Carbidopa 250 mg/ 25 mg. The tablet will be taken with water and in a fasting condition.
  Interventions: Drug: Levodopa 250mg and Carbidopa 25mg Referent Product tablet

INTERVENTIONS:
Drug: Levodopa 250mg and Carbidopa 25mg Test Drug tablet — Investigational Medicinal Product
  Arms: Levodopa and Carbidopa Test Product
Drug: Levodopa 250mg and Carbidopa 25mg Referent Product tablet — Sinemet (Savio Industrial S.R.L, Brazil)
  Arms: Levodopa and Carbidopa Referent Product

SUMMARY:
This study will investigate the bioavailability in fasting male and/or non-pregnant and non- breast feeding female subjects of 1 tablet formulation containing Levodopa 250 mg and Carbidopa 25 mg. The study will be performed at a single site with 44 subjects. Participants will take 1 tablet of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There will be a washout of at least 2 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of Oseltamivir Phosphate 75 mg of 1 capsule formulations with Oseltamivir Phosphate 75 mg and to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Laboratorios Silesia S.A.
* Reference Product: Sinemet [Trademark], product of Savio Industrial S.R.L., Brazil. The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters area under the plasma concentration-time curve from time zero to time t (AUC0 0-t) and from time zero to infinite (AUC0 0-∞), and maximum plasma concentration (Cmax) for total Levodopa and Carbidopa will be determined. Participants will be confined in the study site for approximately 68 hours during the entire study (for 10 hours pre-dosing and for 10 hours post dosing in period II) during which pharmacokinetic (PK) blood samples will be obtained. 23 blood samples will be taken up to 10 hours after the administration in each period. The washout period between the two study periods will be at least 2 days. The samples from each participant will be analyzed with validated LC-MS/MS method for estimation of Levodopa and Carbidopa in plasma. The safety objective is to evaluate the tolerability of both formulations in subjects by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or non-pregnant, non-breast feeding female literate volunteers of 18 to 45 years (both years inclusive) with BMI of 18.50 - 29.99 Kg/m2 and weight > 50 Kg.
2. Healthy volunteers as evaluated by medical history, vitals and general clinical examination.
3. Normal or clinically insignificant biochemical, hematological, urine and serology parameters.
4. Normal or clinically insignificant ECG.
5. Negative urine test for drugs of abuse for both males and females and negative pregnancy test for females and do not plan to become pregnant during course of the study and for 03 months after completion of study.
6. Volunteers who are willing to use acceptable methods of contraception (barrier method/IUD/surgical) or abstinence, for the entire duration of the study and do not plan to be pregnant for at least 1 month after the last drug administration.
7. Volunteers who can give written informed consent and communicate effectively.

Exclusion Criteria:

1. History of any major surgical procedure in the past 03 months.
2. History of any clinically significant cardiac, gastrointestinal, respiratory, hepatic, renal, endocrine, neurological, metabolic, psychiatric and hematological disorders.
3. History of chronic alcoholism/ chronic smoking/ drug of abuse.
4. Volunteers with known hypersensitivity to Levodopa and Carbidopa or any of the excipients.
5. History of consumption of tobacco containing products within 48 hours prior to proposed time of dosing
6. Volunteer who are positive for hepatitis B surface antigen, anti-hepatitis C antibody, treponemal antibodies and human immunodeficiency virus (HIV 1&2) antibodies.
7. Present or past history of intake of drugs or any prescription drug or over the counter (OTC) drugs within 14 days which potentially modify kinetics / dynamics of Levodopa and Carbidopa or any other medication judged to be clinically significant by the investigator.
8. History of consumption of grapefruit and/or its products within 10 days prior to the start of study.
9. Volunteer who had participated in any other clinical study or who had bled during the last 03 months before check-in.
10. History of consumption of one or more of the below, 48 hours prior to dosing: Xanthine containing food or drinks such as cola, chocolate, coffee or tea, citrus fruits or items (lime, lemon and orange), alcohol and any other food/beverage known to have interactions as deemed by the investigator.
11. Volunteers who are dysphagic

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Total Levodopa and Carbidopa: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | 23 samples up to 10 hours will be taken after the administration in each period
Total Levodopa and Carbidopa: area under the plasma concentration-time curve from 0 to time t (AUC0-∞) | 23 samples up to 10 hours will be taken after the administration in each period
Total Levodopa and Carbidopa: Maximum plasma concentration (Cmax) | 23 samples up to 10 hours will be taken after the administration in each period
Total Levodopa and Carbidopa: Time to achieve maximum plasma concentration (tmax) | 23 samples up to 10 hours will be taken after the administration in each period

CONTACTS AND LOCATIONS:
Locations (1):
- Azidus Laboratories Ltd., Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No